CLINICAL TRIAL: NCT04994834
Title: Characterization of the Gastrointestinal Microbiota in Term Newborn Infants After 4 Weeks Supplementation of Probiotics - an Open Label Pilot Study
Brief Title: Characterization of the Gastrointestinal Microbiota in Term Newborn Infants After 4 Weeks Supplementation of Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chr Hansen (Industry)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: ChrHansen (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HND-IN-037
Record Dates: First submitted 2021-06-30; First posted 2021-08-06 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2021-08

CONDITIONS: Gut Microbiota
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Probiotics
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Once a day daily intake of probiotics for at least 28 consecutive starting within 24 hours after birth

SUMMARY:
A mono center, open label, pilot study in term newborn infants. The study will investigate the effect of supplementation with probiotics on the presence of total Bifidobacterium in the infant feces.

DETAILED DESCRIPTION:
The four weeks intervention starts within 24 hours after birth of the study subject and the investigational product will be given for 28 days, followed by a two weeks follow-up period without any intake of the investigational product.

During the entire study period, five visits are scheduled. Visit 2 to Visit 5 are home visits by the study midwife. From Visit 2 and throughout the study period (Visit 2 to Visit 5) the parents will be asked to complete a diary daily.

Infant stool samples will be collected on multiple occasions during the study, as well as maternal breast milk samples, stool and urine samples and samples from vagina. In addition, sample from placenta, umbilical cord, umbilical cord blood and amnion fluid will be collected. Mothers will be asked to complete electronic questionnaires daily during the course of the study.

ELIGIBILITY:
Infants to be enrolled at birth.

Inclusion Criteria for Infants (study subjects)

* Gestational age at birth ≥ 37±0 ≤ weeks 42±0 weeks
* Birthweight more than 2500 g
* No exposure to oral or intravenous antibiotics
* No complications that need medical interventions (e.g. respiratory distress symptoms or infections)
* Both legal guardians provided voluntary written informed consent on behalf of the infant

Pregnant women:

* Women age above 18 years at informed consent
* Singleton pregnancy
* Uncomplicated pregnancy
* No use of medication
* Aim to give birth vaginally and breastfeed
* No use of probiotics during the last month before estimated birth and until six weeks postpartum
* Provided voluntary written informed consent

Exclusion criteria for Infants (study subjects)

• Admission to the neonatal intensive care unit (NICU)

Ages: 0 Days to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Recovery of the investigational product in the infant feces | 28 days after birth
  Presence of the investigational product in infant fecal samples after 4 weeks of supplementation (Visit 4) using PCR

SECONDARY OUTCOMES:
Total fecal Bifidobacterium in infant fecal samples | Baseline, Day14, Day 28
  Total fecal Bifidobacterium in infant fecal samples after 4 weeks supplementation Quantification of total Bifidobacterium will be determined by PCR.
Characterization of the infant intestinal microbiota after 4 weeks supplementation | Baseline, Day 14, Day 28
  Characterization of the infant intestinal microbiota after 4 weeks supplementation of the investigational product using sequencing
Adverse events (Safety) | up to 6 weeks
  Frequency and severity of adverse events

OTHER OUTCOMES:
Mothers fecal microbiota | Baseline
  Characterization of mother's microbiota from fecal samples will be assessed using sequencing to examine the microbiota for similarities with the infant
Infant Gastrointestinal Problems | 42 days
  Infant Gastrointestinal Problems will be measured using ROME IV Diagnostic Questionnaires for Pediatric Functional Gastrointestinal Disorders for Neonates and Toddlers: Parent-Report Form for Neonates Section A - Infant Gastrointestinal Problems
Stool frequency and consistency | 42 days
  Infant stool frequency and consistency will be measured using Amsterdam Stool Chart.
Reflux | 42 days
  Reflux will be measured using Infant Gastroesophageal Reflux Questionnaire Revised (I-GERQ-R)
Breastmilk microbiome | Baseline, Day 14, Day 28
  Microbiome of the breastmilk to be assessed using sequencing to explore a potential microbiota of the breastmilk
Mothers vaginal microbiota | Baseline
  Characterization of mother's vaginal microbiota will be assessed using sequencing to examine the microbiota for similarities with the infant

CONTACTS AND LOCATIONS:
Overall Officials: Lars Henning Pedersen, Professor, Principal Investigator — Department of Gynecology and Obstetrics, Aarhus University Hospital
Locations (1):
- Department of Gynaecology and Obstetrics, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
To share IPD not decided yet